CLINICAL TRIAL: NCT01484743
Title: Nationwide Prospective Study of Surgical Risk Factors for Poor Outcome After Parastomal Hernia Repair
Brief Title: Risk Factors for Morbidity After Parastomal Hernia Repair
Acronym: PAHEREP
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: Parastoma
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Parastomal Hernia
Keywords: recurrence; readmission; reoperation; mortality; morbidity
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with parastomal hernia repair: Patients registered in the Danish Ventral Hernia database
  Interventions: Procedure: differences in surgical techniques

INTERVENTIONS:
Procedure: differences in surgical techniques — follow the risk for morbidity after incisional hernia repair

SUMMARY:
The Danish Ventral Hernia Database (DVHD) registers 37 different perioperative parameters. The aim of present study is to use large-scale data from DVHD to uncover risk factors for readmission, reoperation (any indication), death and reoperation for recurrence after parastomal hernia repair.

DETAILED DESCRIPTION:
All principal parastomal hernias registered in the Danish Ventral Hernia Database are included in the study. The included patients will be followed in up to 4 years in order to identify correlation between technical aspects of the hernia repair and postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* All parastomal hernia repairs registered in the Danish National Ventral Hernia Database

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All incisional hernia repairs registered in the Danish National Hernia Database from January 1st 2007 to December 31st 2010
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Recurrence repair | up to 4 years after operation
  Surgical risk factors for recurrence repair after parastomal hernia repair.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Helgstrand, MD, Principal Investigator — Dept. surgery Koege hospital
Locations (1):
- Køge Hospital, Køge, Region Sjælland, Denmark